CLINICAL TRIAL: NCT06098547
Title: LIver Transplantation for Non-Resectable Intrahepatic CholAngiocarcinoma (LIRICA)
Acronym: LIRICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Ospedaliera (Other)
Collaborators: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Principal Investigator, Enrico Gringeri, Associate Professor, Azienda Ospedaliera di Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOP 3006; LIRICA (Other: University of Padova)
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Liver transplantation
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Experimental): Candidates will be evaluated by theMultidisciplinary Group after routine radiological studies (CT, MRI, PET-MR/CT).
  Patients will receive 6 months of standard of care chemotherapy and undergo PET-MR with FDG to exclude the presence of extrahepatic disease.
  Following completion of therapy, patients will undergo radiological restaging. If the disease is resectable, the patient will be considered for curative-intent surgical resection; if not, the patients will be evaluated by the Center's Multidisciplinary Transplantation Group.
  Patients will continue chemotherapy until a compatible liver becomes available. If there are no further contraindications, exploratory laparotomy and surgical nodal staging of the tumor will be performed at the time of transplantation. If there are no signs of extrahepatic disease, transplantation will be conducted according to institutional protocols.
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Patients will undergo liver transplantation according to the standard procedures of the institutional Center's protocol (cadaveric or living donor transplantation, whole or partial liver).
  Liver transplantation is preceded by an exploratory laparotomy with clinical evaluation and frozen section examination of lymph nodes in the hepatoduodenal ligament and along the common hepatic artery/celiac axis.

SUMMARY:
LIRICA is a prospective non-randomized study aimed at exploring the outcome of liver transplantation in selected patients with unresectable iCCA after a downstaging/disease control protocol with standard of care chemotherapy, in terms of overall survival and quality of life. Additionally, the study aims to identify pre-transplant biological markers and clinical factors that can stratify patients with the best post-transplant prognosis. Finally, the study aims to investigate the role of preoperative PET-MR, especially in relation to lymph node locations, by correlating the results with histological examination after iliac lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of iCCA
* First diagnosis of iCCA
* Recurrence after R0 hepatic resection, N0, M0 without macrovascular invasion
* Disease considered unsuitable for hepatic resection based on tumor location and extent or underlying liver dysfunction
* Absence of major vascular invasion, extrahepatic disease, or involvement of regional lymph nodes detected on radiological study
* No evidence of extrahepatic metastatic disease after chest-abdomen-pelvis CT and PET-MR (or PET-CT)
* At least six months have passed since the first diagnosis of iCCA (or recurrence) to the date of inclusion on the liver transplant waiting list
* The patient has received at least six months of SOC chemotherapy, achieving disease stability or partial response (according to RECIST version 1.1) at the time of listing for transplantation
* Hematochemical evaluation: Hb ≥ 9 g/dL, Leukocytes ≥ 3.0 X 109/L, Neutrophils ≥ 1.5 X 109/L, Platelets ≥ 100,000/mm3 (≥ 10 X 109/L), Total Bilirubin ≤ 3 mg/dL (≤ 51 umol/L), AST or ALT ≤ 5 times the upper limit of normal, Serum Creatinine and Urea < 1.5 times the upper limit of normal
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 1
* Patient's BMI ≥ 18 and ≤ 30 kg/m2
* Signed informed consent, and expected patient cooperation for treatment and follow-up, must be obtained and documented according to good clinical practice and national/local regulations

Exclusion Criteria:

* Tumor involving nearby extrahepatic structures (including involvement of major hepatic vessels) by direct invasion (T4 per AJCC 8th edition)
* Tumor penetrating the visceral peritoneum (T3 per AJCC 8th edition)
* Previous extrahepatic metastatic disease
* Prior neoplasms, except those treated curatively for more than 5 years without recurrence
* Known history of human immunodeficiency virus (HIV) infection
* Known history of solid organ or bone marrow transplantation
* Substance abuse and medical, psychological, or social conditions that may interfere with the patient's participation in the study or with the evaluation of study outcomes
* Pregnant or breastfeeding women
* Medical-surgical contraindications for liver transplantation
* Any reason for which, in the investigator's judgment, the patient should not participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 and 5 years
  Survival from time of transplantation to time of death or last follow up

SECONDARY OUTCOMES:
OS comparison with chemotherapy alone | 3 years
  Comparison of 3-year survival between patients enrolled in the LIRICA study and survival of a population balanced for prognostic factors and disease characteristics from the database of the Veneto Oncological Institute (IOV)
Disease-Free Survival (DFS) | 3 and 5 years
  Survival from time of transplantation to time of death or first evidence of recurrence fo disease
Overall survival from the time of recurrence | 5 years
  Survival from time of recurrence to time of death or last follow up
PFS comparison with chemotherapy alone | 3 years
  Comparison of 3-year Progression-Free Survival (PFS) between the per-protocol population of patients enrolled in the LIRICA study and the PFS of the population from the Veneto Oncological Institute (IOV) database
Biological markers | 5 years
  Correlation of overall survival and recurrence with tissue and circulating biological markers (immunohistochemistry, proteomics, circulating tumor cells, circulating tumor DNA, new molecular markers)
Morbidity | 90 days
  Morbidity at 90 days (according to Clavien-Dindo and Comprehensive Complication Index, CCI)
Cancer-related mortality | 3 and 5 years
  Risk of mortality with sole relation to death by tumor progression and
Drop out | 5 years
  Percentage of patients who do not complete the procedure (drop-out) stratified by cause
Concordance of surgical and PET_RM staging (number, size, location) | Perioperative
  Asses if suspicious lymph nodes described at the preoperative PET-RM confirm to be pathological at the histological evaluation after lymphadenectomy of the hepatic hilum and exploratory laparotomy. Lymph nodes will we evaluated by number, size and location
Quality of life assessed using EORTC QLQ-C30 | 5 years
  Quality of life assessed using EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer QLG Core Questionnaire) 30 items questionnaire (scale 1-4 or 1-7, 1 being the lowest and 4 or 7 the highest, accordingly)
Quality of life assessed using FACT-Hep questionnaire | 5 years
  Quality of life assessed using FACT-Hep questionnaire (Functional Assessment of Cancer Therapy - Hepatobiliary) questionnaire about quality of life in the last 7 days (scale 0-4, 0 being the lowest and 4 the highest)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Gringeri, Prof., Principal Investigator — Azienda Ospedale Università di Padova
Locations (1):
- Azienda Ospedale Università di Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No